CLINICAL TRIAL: NCT07216573
Title: Continuous Blood Pressure Monitoring During Outpatient Surgery
Brief Title: The Continuity Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2025-06
Record Dates: First submitted 2025-09-19; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1 - Standard of Care (Experimental): Study device data are blinded to the provider
  Interventions: Device: HemoSphere Vita Monitor, VitaWave or VitaWave Plus Finger Cuff Adult, ForeSight Large Sensors
- Cohort 2 - Standard of Care with cNIBP Monitoring (Experimental): Study device continuous non-invasive blood pressure data are unblinded to the provider
  Interventions: Device: HemoSphere Vita Monitor, VitaWave or VitaWave Plus Finger Cuff Adult, ForeSight Large Sensors

INTERVENTIONS:
Device: HemoSphere Vita Monitor, VitaWave or VitaWave Plus Finger Cuff Adult, ForeSight Large Sensors — Devices are applied for monitoring throughout the duration of the procedure.

SUMMARY:
A before & after interventional cohort study comparing intermittent blood pressure measurement using the oscillometric arm cuff to continuous noninvasive blood pressure measurement using the VitaWave finger cuffs in subjects undergoing elective surgery in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 18 years
3. ASA Physical Status ≥ 2
4. Scheduled for elective noncardiac surgery with intermittent arterial blood pressure monitoring using oscillometric arm cuff

Exclusion Criteria:

1. Patient who is known to be pregnant
2. Patient with existing or planned arterial pressure catheter
3. Patient in whom systolic arterial pressure differs by more than 20 mmHg between the right and left arms
4. Inability to place oscillometric cuff on the subject's upper extremity
5. Extreme contraction of the smooth muscle in the arteries and arterioles of the lower arm and hand, such as may be present in patients with Raynaud's disease
6. Finger or hand deformity that prevents proper placement of finger cuff by visual inspection
7. Inability to place finger cuffs due to subject anatomy, condition, or obstructive paraphernalia (such as false nails)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of adult patients undergoing elective noncardiac surgery in the outpatient setting who experience hypotension, defined as a MAP < 65 mmHg, for a total duration of at least 5 minutes. | Through Study Completion, approximately 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No